CLINICAL TRIAL: NCT02437994
Title: Impact of a Pulmonary Rehabilitation Program on the PROactive Tool
Brief Title: Pulmonary Rehabilitation Program and PROactive Tool
Acronym: PROactive
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Thorax Research Foundation (Other)
Responsible Party: Principal Investigator, IOANNIS VOGIATZIS, Principal Invetsigator, Thorax Research Foundation
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 933
Record Dates: First submitted 2015-04-21; First posted 2015-05-08 (Estimated); Last update posted 2016-05-06 (Estimated); Status verified 2016-05

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pulmonary Rehabilitation (Experimental): The rehabilitation program will be multidisciplinary and will include supervised exercise training (interval exercise and resistance exercises), breathing control and relaxation techniques, methods of clearance of pulmonary secretions, disease education, dietary advice, and psychological support on issues relating to chronic disability.
  Interventions: Behavioral: Pulmonary Rehabilitation
- Control (No Intervention): In addition, a control group (Group C) which will not participate in the rehabilitation program (usual care) will be include at the same time as patients in Group A and B so as to be able and independently address study objectives 2 and 3 and 4. Group C will also randomized to those into paper-pencil version and electronic version.

INTERVENTIONS:
Behavioral: Pulmonary Rehabilitation — The rehabilitation program will be multidisciplinary and will include mandatory supervised exercise training at appropriate training intensity, other components of the program can be breathing control and relaxation techniques, methods of clearance of pulmonary secretions, disease education, dietary advice, and psychological support on issues relating to chronic disability. Six minute walking tests, and improvements in dyspnea sensation (CRDQ) will be used to benchmark the effect of a program provided by a given team.
  Arms: Pulmonary Rehabilitation

SUMMARY:
Pulmonary rehabilitation is an essential non pharmacological treatment option which reduces dyspnea sensations, increase exercise tolerance, improves health related quality of life and reduces the burden on health care resources (1). Pulmonary rehabilitation is likely an ideal intervention to validate the PROactive tool as responses to pulmonary rehabilitation are clinically significant in terms of exercise tolerance and particularly activity related symptoms. Nevertheless, the response to pulmonary rehabilitation is variable and about one out of three patients does not present a clinically important response. Pulmonary rehabilitation may therefore be an intervention that allows studying the conceptual model around the PROactive tools, anchoring the new PROs (Patient Report Outcome) to outcomes that are well known to change with rehabilitation: exercise induced symptoms, functional exercise tolerance and health related quality of life.

Study objectives

Main objectives

A primary aim is to test reliability of the paper-pencil versus the electronic scoring version of the PROactive tool in terms of assessing the effect of pulmonary rehabilitation on the components of the PROactive tool and on the mode of administration.

The secondary aim of the proposed project is to investigate the effects of a multidisciplinary outpatient hospital-based, pulmonary rehabilitation program on: i) daily physical activity (number of daily steps, vector magnitude unit and movement intensity and ii) the components of the Proactive tool.

Additional study objectives

A third aim of this project is to investigate whether the magnitude of change in daily physical activity and the components of the PROactive tool in general is associated with the magnitude of changes in frequently used rehabilitation related end-points including, functional capacity, exercise capacity and health-related quality of life following the completion of a comprehensive pulmonary rehabilitation program.

A forth aim of this project is to investigate whether the magnitude of change in daily physical activity and the components of the PROactive tool in general is associated with the magnitude of changes in physiological indices including cardiovascular and respiratory adaptations following completion of a comprehensive pulmonary rehabilitation program.

DETAILED DESCRIPTION:
Study hypotheses

The patients involved during Work Package 4 of the PROactive Project showed a good conformity with the use of electronic devices such as the electronic version of the PROactive tool. As the paper-pencil version is anticipated to be equally easy to manage from the patients as the electronic version, therefore it is expected an excellent agreement between the paper-pencil and the electronic version in terms of assessing the effect of pulmonary rehabilitation on the components of the PROactive tool.

A pulmonary rehabilitation program of at least 8-10 weeks is considered sufficient to induce reduction in daily and exercise induced symptoms, improvements in functional capacity and exercise tolerance and increase in health related quality of life in patients with COPD. Since low levels of physical activity are associated with reduced exercise performance and increased daily symptoms, it is anticipated a significant improvements in daily physical activity levels (as measured by daily number of steps, vector magnitude unit and movement intensity) and in the components of the Pro-Active tool following the completion of the pulmonary rehabilitation program.

Recent published studies funded form PROactive Project revealed that activity monitoring outputs are associated with the cardiovascular, respiratory, and metabolic load of exercise in COPD patients. Therefore it is expected to found significant associations between daily physical activity levels and the components of the PROactive tool in general with functional capacity, exercise capacity and cardio-respiratory adaptations following completion of a comprehensive pulmonary rehabilitation program.

Study population

A convenience sample of clinically stable patients with COPD will be recruited from the academic centers' Outpatient Clinic on the following entry criteria: 1) a post-bronchodilator forced expiratory volume in one second (FEV1) <70% predicted without significant reversibility (<12% change of the initial FEV1 value or <200 ml) and 2) optimal medical therapy according to Global Initiative for Chronic Obstructive Lung Disease (GOLD) (2). Exclusion criteria will include: 1) Orthopedic, neurological, and other musculoskeletal complaints that could impair normal movement patterns, 2) respiratory diseases other than COPD (e.g. asthma), 3) hospital admission or COPD exacerbations within the previous 4 weeks 4) patients not on optimal pharmacotherapy. The study will be approved by the University Hospital Ethics Committee and the PROactive EC and patients will provide informed written consent.

Study Design

The total number of patients will be automatically assigned in two groups: Group A will consist of patients who will score only the paper-pencil version of the clinical visit version of PROactive tool. Group B will consist of patients who will score only the electronic version of the clinical visit version of PROactive tool. Randomization should be stratified by site. In addition, a control group (Group C) which will not participate in the rehabilitation program will be include at the same time as patients in Group A and B so as to be able and independently address study objectives 2 and 3 and 4. Group C will also randomized to those into pape-pencil version and electronic version.

Following completion of the first week (i.e.: V1) patients will complete a multidisciplinary pulmonary rehabilitation program. Following completion of the rehabilitation program patients will perform one more visit (V2). During visit 1 and 2 patients will perform the measurements indicated in tab

Rehabilitation program

The rehabilitation program will be multidisciplinary and will include mandatory supervised exercise training at appropriate training intensity, other components of the program can be breathing control and relaxation techniques, methods of clearance of pulmonary secretions, disease education, dietary advice, and psychological support on issues relating to chronic disability. Six minute walking tests, and improvements in dyspnea sensation (CRDQ) will be used to benchmark the effect of a program provided by a given team.

Data management

Patient data will be stored in a randomized database as for WP2D. Data will be analyzed centrally and the relevant PRO data and accessory end points will be available in a format to allow integration with other PROactive WP6 studies.

Assessments

Primary outcomes

PROactive tool

Physical activity measurements in terms of daily number of steps and vector magnitude unit (VMU) will be performed primarily by the ''Actigraph'' triaxial activity monitor whilst patients will answer to the clinical visit questionaire of Proactive tool as well as to the PROactive questionnaires (i.e. CCQ, CRQ, HADS, CAT, SGRQ). Additionally, in a subgroup of patients assigned in each of the three groups (i.e. Group A, B, C) activity monitoring measurements in terms of walking intensity will be performed by the Minimod (McRoberts BV) activity monitor.

Secondary outcomes

Anthropometrics-Body composition

Body weight will be measured to the nearest 0.1 kg with a digital scale and height will be measured to the nearest 0.5 cm with a stadiometer. Body mass index (BMI) will be calculated as the ratio of weight (in kilograms) to height (in metres) squared. Body composition will be estimated by a bioelectric impedance device.

Recording data:

Recording the following parameters: weight, height, total body water, fat mass (FM), fat free mass (FFM).

Lung function

Spirometry, body plethysmography and single breath transfer factor for carbon dioxide will be measured according to the American Thoracic Society/European Respiratory Society standards after administering 400μg salbutamol (3). Post bronchodilator static lung volumes will be assessed using a body-box (whole body plethysmography).

Recording data:

Recording the following parameters: FEV1 and FVC, TLC, RV, TGV and TLco.

Exercise capacity

Incremental exercise test

The incremental exercise test will be performed on an electromagnetically braked cycle ergometer (Ergoline 800; Sensor Medics, Anaheim, CA, USA) with a ramp increase of load increments of 5 to 25 Watt/min until the patient reaches volitional exhaustion.

Recording data:

Recording the following parameters: peak work rate, peak oxygen uptake, peak heart rate, minute ventilation at Iso-Work and peak minute ventilation, SpO2, dyspnea sensation and leg discomfort (10-Borg scale).

Six-minute walking test

The 6-minute walk test (6MWT) will be measured following the instructions of the American Thoracic Society (ATS) recommendations.

Recording data:

Before and after exercise test: heart rate, SpO2, dyspnea sensation and leg discomfort (10-Borg scale) and distance walked.

Skeletal muscle function test

Patients will be studied seated in the quads chair, with hip and knee flexion of 90 degrees. An inextensible strap will be placed around the ankle, immediately proximal to the malleoli, adjusted to ensure the knee remains at 90 degrees flexion. The ankle strap will be connected to a strain gauge mounted on the back of the chair, and runs perpendicular to both the ankle and the strain gauge. A seatbelt will be secured across the subject's hips to stabilize the pelvis

Recording data:

Record the following parameters: strength expressed in kg and leg length.

Central hemodynamics

Cardiac output will be measured non-invasively throughout the incremental exercise test on the treadmill using a portable impedance cardiography device (PhysioFlow , Manatec Biomedical, France) (4).

Recording data:

Cardiac output, heart rate and stroke volume will be recorded continuously at rest, during exercise and recovery throughout the tests.

Statistical analysis and randomization

Baseline characteristics, including age, gender, as well as clinical and functional data, including but not limited to lung function, body composition, quadriceps strength, 6MWT, CRQ, CCQ, HADS, CAT, SGRQ and PROactive monitors outputs, will be summarized according to number and percentage for qualitative variables, mean and standard deviation for quantitative variables with normal distribution, and median and 25th-75th percentiles for quantitative variables with non-normal distribution. The effectiveness of the rehabilitation program between and within groups on daily physical activity levels and PROactive tool will be tested using an analysis of variance (ANOVA) model. Pearson correlation coefficient analysis will be performed to determine the relationship between variables using as a dependent variable the physical activity levels and PROactive tool score while the independent variables included functional capacity, exercise capacity, PROactive questionnaires, metabolic, respiratory, central hemodynamic parameters that were measured following the completion of the rehabilitation program.

Randomization Stratified randomization will be applied taking into account patient's baseline daily physical activity levels, namely weekly median steps.

ELIGIBILITY:
Inclusion Criteria:

Clinically stable patients with COPD will be recruited from the academic centers' Outpatient Clinic on the following entry criteria:

1. a post-bronchodilator forced expiratory volume in one second (FEV1) <70% predicted without significant reversibility (<12% change of the initial FEV1 value or <200 ml) and
2. optimal medical therapy according to Global Initiative for Chronic Obstructive Lung Disease (GOLD) (6).

Exclusion Criteria:

1. Orthopedic, neurological, and other musculoskeletal complaints that could impair normal movement patterns,
2. respiratory diseases other than COPD (e.g. asthma),
3. hospital admission or COPD exacerbations within the previous 4 weeks
4. patients not on optimal pharmacotherapy.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2013-10; Primary Completion 2016-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Proactive tool (clinical visit version) | 7 days
  Proactive tool is a patient-reported outcome which combines a 12-item self-administrated questionnaire and activity monitor score in order to assess daily physical activity in patients with COPD. Proactive tool can be scored as a simple sum of the scores of the items (each item can be scored mostly from 0 to 4), with lower scores indicating poorer physical activity.

SECONDARY OUTCOMES:
Daily Physical activity as measured by a validated for COPD patients triaxial accelerometers | 7 days
  Daily physical activity in terms of daily number of steps, vector magnitude units (VMU) per activity minute and walking intensity.

CONTACTS AND LOCATIONS:
Overall Officials: CHARALAMBOS ROUSSOS, PhD, MD, Study Director — Thorax Research Foundation
Locations (1):
- Pulmonary Rehabilitation Centre, Sotiria Hospital, 1st Departments of Respiratory Medicine, National and Kapodistrian University of Athens, Athens, Greece

REFERENCES:
- [Background] 1. Nici L. American Thoracic Society/ Respiratory Society statement of pulmonary rehabilitation. American Journal Respiratory Critical Care Medicine 173: 1390-1413, 2006. 2. Global Initiative for Chronic Obstructive Lung Disease. Global strategy for the diagnosis, management, and prevention of chronic obstructive pulmonary disease. Executive summary. 2005 3. Rabe K.F. Global strategy for the diagnosis, management, and prevention of chronic obstructive pulmonary disease: GOLD executive summary. American Journal Respiratory Critical Care Medicine 176: 532-555, 2007. 4. Charloux A. Exercise by a new impedance cardiography device: comparison with the direct Fick method. European of Applied Physiology 82: 313-320, 2000.
- [Derived] Louvaris Z, Spetsioti S, Kortianou EA, Vasilopoulou M, Nasis I, Kaltsakas G, Koulouris NG, Vogiatzis I. Interval training induces clinically meaningful effects in daily activity levels in COPD. Eur Respir J. 2016 Aug;48(2):567-70. doi: 10.1183/13993003.00679-2016. Epub 2016 Jun 23. No abstract available. PMID 27338191
- See also: Thorax Research Foundation — http://www.thorax.org.gr/index.php/en/the-foundation/and/